CLINICAL TRIAL: NCT06132633
Title: A Pilot Study for the Adaptation of Neospot Device for Health Care Among Out-Patients at Primary Health Facilities in Nairobi and Kajiado Counties, Kenya
Brief Title: A Pilot Study for Adaptation of Neospot Device for Health Care at Primary Health Facilities in Kenya
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neopenda, PBC (Industry)
Collaborators: Amref Health Africa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P1339/2023
Record Dates: First submitted 2023-09-07; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Morbidity
Keywords: Morbidity; Vitals Measurement; Health

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional study design. All participants receive the same intervention of our Neospot vitals measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neospot Vitals Measurement (Experimental): Neospot is a 5-in-1 wearable vitals measurement device designed to measure temperature, blood pressure, pulse rate, respiratory rate and blood oxygen saturation. For the standard of care vitals measurement, conventional vital signs will be measured using mercury blood pressure cuffs and infrared or mercury thermometers for blood pressure and temperature respectively, pulse oximeter for oxygen saturation and a 1-minute count of heart rate and breathing rate.
  Interventions: Device: Neospot vitals measurement

INTERVENTIONS:
Device: Neospot vitals measurement — Vitals of participants in the intervention group will be measured using neospot alongside standard of care measurement.

SUMMARY:
Neospot device is a 5-in-1 wearable vital signs monitor designed to measure temperature, blood pressure, pulse rate (PR), respiratory rate (RR) and blood oxygen saturation (SPO2). We propose to study the experiences of patients and nurses regarding spot measurement of vital signs at the outpatient department in primary care facilities in Kenya. The study aims to investigate the capability, opportunity, and motivation of nurses to use the Neospot device for vital signs measurement in level 3 facilities in Kenya by validating the accuracy of the Neospot and assessing the experience of patients while using the Neospot, the study also aims to assess the experiences of nurses as they use the Neospot and determine how the Neospot affects their workflow.

DETAILED DESCRIPTION:
This study intends to investigate the experiences of both nurses and patients in the use of a specific brand of such a device known as the 'neospot' device in various sub county, health centres in Kenya. The study also aims at finding out whether the device affects the rate and efficiency of how nurses work in these facilities.

The study will apply a cross sectional design, three facilities will be used as the sampling frame two urban facilities from Nairobi County and one peri urban rural facility from Kajiado county. The participants will be selected randomly. Data will be obtained from a total of 159 randomly selected patients, all the nurses who will be on duty will also be included as participants in the study and the team leaders will be interviewed as key informants for qualitative data. Quantitative data will be analysed using SPSS version 24 for descriptive and inferential statistics, NVIVO software will be used to analyse the qualitative data to determine the themes. Study Duration: Data collection, analysis and report writing will take 4 ½ months.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 70 years of age
* In stable condition
* Willing to give consent to participate in the study

Exclusion Criteria:

* Very ill and unstable patients who need emergency care
* Patients with medical conditions that are characterized by rapid changes in vital signs such as thyroid disorders
* Patients who have skin lesions on the forehead where the device is to be fixed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Capability, opportunity and motivation of nurses to use the Neospot device for vital signs measurement | From enrolment, monitoring, data extraction and analysis over a period of 4 months
  Number of nurses reporting positive experiences and improved workflow as a result of utilizing the neospot product as responded in surveys

SECONDARY OUTCOMES:
Accuracy of vitals measurement of Neospot device compared to traditional equipment | From enrolment, monitoring, data extraction and analysis over a period of 4 months
  We want to validate the accuracy of the Neospot device to measure temperature, SPO2, pulse rate and respiratory rate by comparing similarities and differences to the traditional devices vital signs readings
Experiences of patients using the Neospot vitals measurement device | From enrolment, monitoring, data extraction and analysis over a period of 4 months
  Number of patients reporting positive experience with our Neospot device through surveys
Acceptability of Neospot device by nurses for adoption in health facilities | From enrolment, monitoring, data extraction and analysis over a period of 4 months
  Number of nurses willingness to adopt the use the Neospot device as their primary vital sign measurement tool post utilization, determined through surveys
Effects of Neospot vitals measurement device on nurses' workflow | From enrolment, monitoring, data extraction and analysis over a period of 4 months
  Number of nurses reporting positive impact of the Neospot device on efficiency and improved workflow through surveys

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Oyieke, Principal Investigator — Amref International University
Locations (1):
- Langata, Kianda 42 and Matasia Health Centre, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No